CLINICAL TRIAL: NCT06152042
Title: Phase 2 Randomized, Double-blind Trial of BMF-219 Compared to Placebo in Participants With Type 1 Diabetes Mellitus
Brief Title: Phase 2 Trial of BMF-219 in Participants With Type 1 Diabetes Mellitus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor made a business decision to terminate the study based on prioritization of portfolio.
Sponsor: Biomea Fusion Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COVALENT-112
Record Dates: First submitted 2023-11-10; First posted 2023-11-30 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: COVALENT-112 consists of two parts. Part 1 is a single-arm, open-label study; Part 2 is a randomized, double-blind, placebo-controlled study. Both will enroll adults with Stage 3 T1D (HbA1c ≥6.5 and ≤ 10.0%).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): Part 1 uses a randomized, open-label design with parallel assignment between 2 treatment arms in each cohort. The Part 1 Eligible participants will be randomly assigned by cohort to 1 of 2 treatment arms:
  * Cohort 1: Participants with T1D diagnosed within 3 years with C-peptide concentration ≥0.2 nmol/L
  * Arm A: BMF-219 100 mg QD for 12 weeks
  * Arm B: BMF-219 200 mg QD for 12 weeks
  * Cohort 2: Participants with T1D diagnosed between 3 to 15 years with C-peptide concentration ≥0.08 nmol/L.
  * Arm A: BMF-219 100 mg QD for 12 weeks
  * Arm B: BMF-219 200 mg QD for 12 weeks
  Interventions: Drug: BMF-219
- Part 2 (Experimental): Part 2
  Part 2 uses a randomized, double-blind, placebo-controlled design with parallel assignment among 3 treatment arms. Eligible participants will be randomly assigned to 1 of 3 arms using a 1:1:1 ratio:
  * Arm A: BMF-219 100 mg QD for 12 weeks
  * Arm B: BMF-219 200 mg QD for 12 weeks
  Interventions: Drug: BMF-219
- Placebo Comparator (Placebo Comparator): Part 2 Study Double Blind Arm C matching placebo for 12 weeks.
  Interventions: Drug: BMF-219

INTERVENTIONS:
Drug: BMF-219 — BMF-219 is an orally bioavailable, covalent small-molecule menin inhibitor.

SUMMARY:
Phase 2 Trial of BMF-219 in Participants with Type 1 Diabetes Mellitus.

DETAILED DESCRIPTION:
Study COVALENT-112 is a 52-week, Phase 2 trial designed to examine beta-cell function, insulin sensitivity, and both glucose and lipid metabolism in participants with T1D treated with BMF-219. BMF-219 is an orally bioavailable, covalent small-molecule menin inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, age ≥18 and ≤70 years.
2. Diagnosed with stage 3 T1D within the following timeframes:

   * Part 1 Cohort 1: Participants diagnosed within 3 years prior to screening.
   * Part 1 Cohort 2: Participants diagnosed between 3 to 15 years prior to screening
   * Part 2 : Participants diagnosed within 15 years prior to screening.
3. Treated with insulin only for at least 2 months prior to screening and proficient in the following in the opinion of the investigator:

   * Counting carbohydrates
   * Adjusting meal and correction boluses based on glucose readings with a stable insulin/carbohydrate ratio as well as correction factors
   * Adjusting insulin and dietary therapy during special situations (eg, exercise, stress, intermittent diseases)
4. HbA1c ≥6.5 and ≤10.0% at screening.
5. Fasting or stimulated C-peptide Concentration at Screening as follows:

   * C-peptide concentration ≥0.2 nmol/L if diagnosed within 3 years prior to screening.
   * C-peptide concentration ≥0.08 nmol/L if diagnosed between 3 and 15 years prior to screening.
6. Documented history of at least 1 T1D1-related autoantibody.
7. If treated with lipid-lowering therapy, the dose must be stable for at least 30 days prior to screening.
8. Men and women of childbearing potential must use adequate birth control measures for the duration of the trial and at least 90 days after discontinuing study treatment.
9. Women who are not pregnant or lactating.

Exclusion Criteria:

1. Diagnosis of MODY, T2D or any other subtype of diabetes mellitus other than T1D.
2. Have had recurrence (≥2 episodes) of severe hypoglycemia
3. Known self or family history (first-degree relative) of multiple endocrine neoplasia Type 1.
4. Use of diabetes medications except insulin within 2 months prior to screening.
5. Any significant cardiovascular disease or QTcF prolongation within the last 6 months prior to screening.
6. Participants with fasting triglyceride ≥500 mg/dL.
7. Have an eGFR <60 mL/min/1.73 m2 by the CKDEPI Creatinine Equation at screening.
8. Impaired liver function, defined as screening AST or ALT >1.5 × ULN, Total bilirubin >1.5 × ULN with the exception of Gilbert's Syndrome.
9. History of acute or chronic pancreatitis, complete pancreatectomy or pancreas transplants.
10. Serum lipase and/or amylase above 1.5 x ULN.
11. Known positive test for HIV, HBV surface antigen and COVID-19.
12. Diagnosis of, or treatment for, any cancer within the last 2 years with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ, melanoma in situ) treated with potentially curative therapy.
13. Active (symptomatic) celiac disease.
14. History of stomach or intestinal surgery that would potentially alter absorption and/or excretion of orally administered drugs.
15. History of cirrhosis.
16. Currently participating in a formal weight loss program and/or are currently using any drugs for weight management within 2 months of screening.
17. Use of Proton pump inhibitors (PPIs) is prohibited.
18. Treatment with a moderate or strong CYP3A4 inhibitor, inducer, or substrate within a week prior to dosing on Day 1.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-12-28 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
To assess the effect on endogenous insulin secretion | 26 Weeks
  Mean change from baseline in stimulated C-peptide AUC.

SECONDARY OUTCOMES:
To assess the effect on endogenous insulin secretion | 26 Weeks
  Maximum stimulated C-peptide: the highest value at any time point during the 4-hour MMTT.
To assess the effect on additional glycemic parameters | 26 Weeks of treatment
  Mean change from baseline in HbA1c.
To assess the effect on additional glycemic parameters | 26 Weeks
  Mean change from baseline in FPG.
To assess hypoglycemia events | 26 weeks
  Percentage of participants with hypoglycemic episodes (with confirmed self-plasma glucose monitoring) including level 2 hypoglycemic events (<54 mg/dL regardless of symptoms) and level 3 (severe) hypoglycemia across different timepoints.
To assess the effect on insulin doses | 26 Weeks
  Change from baseline in mean daily insulin dosing.
Rate of symptomatic hypoglycemic episodes | 26 Weeks and during study duration
  Evaluation and comparison of the number of symptomatic (both minor and severe) hypoglycemic episodes with BMF-219 vs placebo during the study.
Incidence of adverse events | 26 Weeks and during study duration
  Evaluation and comparison of the number of adverse events with BMF-219 vs placebo during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Pablo Frias, MD, Study Director — Biomea Fusion Inc.
Locations (11):
- United States (9):
  - Oceanic Research Group, North Miami Beach, Florida
  - Lucas Research, Inc., Morehead City, North Carolina
  - Alliance for Multispecialty Research, LLC., Norman, Oklahoma
  - University Diabetes & Endocrine Consultants, Chattanooga, Tennessee
  - Velocity Clinical Research, Dallas, Texas
  - Texas Diabetes & Endocrinology, Round Rock, Texas
  - Diabetes & Glandular Disease Clinic, P.A., San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Manassas Clinical Research Center, Manassas, Virginia
- Canada (2):
  - Dr. T.G Elliott Inc. dba BC Diabetes, Vancouver, British Columbia
  - Centricity Research, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No